CLINICAL TRIAL: NCT00924820
Title: A Pilot Study of Systemically Administered Bevacizumab in Patients With Neoplastic Meningitis (NM)
Brief Title: A Pilot Study of Bevacizumab for Neoplastic Meningitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0122; NCI-2009-01610 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-06-18; First posted 2009-06-19 (Estimated); Results first posted 2020-12-31 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Neoplastic Meningitis
Keywords: Neoplastic Meningitis; NM; Advanced Cancers; Brain Cancer; Advanced Cancer; Brain Diseases; Central Nervous System Disorders; CNS; Bevacizumab; Avastin; Anti-VEGF monoclonal antibody; rhuMAb-VEGF; Spinal Cord; meninges; cerebrospinal fluid; CSF
MeSH Terms: conditions — Meningeal Carcinomatosis; Brain Neoplasms; Brain Diseases; Central Nervous System Diseases | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bevacizumab (Experimental): Bevacizumab 10 mg/kg by vein over about 1 hour, every 2 weeks.
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — 10 mg/kg by vein over about 1 hour, every 2 weeks.
  Other Names: Avastin; Anti-VEGF monoclonal antibody; rhuMAb-VEGF

SUMMARY:
The goal of this clinical research study is to learn if and how Avastin (bevacizumab) may affect cancer that has spread to the meninges of the brain or the spinal cord. The safety of this drug will also be studied.

Objectives:

1. Primary:

1. Determine preliminary response data of intravenous bevacizumab in patients with NM

a. As measured by clearance of malignant cells from the Cerebrospinal fluid (CSF) at 2, 4, 6, 12, 18, and 24 weeks, then every 8 weeks up to 54 weeks, and

b. Time to neurological progression (TTNP)

2. Secondary:

1. Evaluate the safety of intravenous bevacizumab in patients with NM
2. Further describe the efficacy of this intervention as measured by

   1. improvement of MR imaging evidence of disease
   2. overall survival
   3. maintenance of quality of life
3. Determine effects of systemically administered bevacizumab on CSF, serum, and urine Vascular endothelial growth factor (VEGF)levels levels
4. Correlate changes in CSF VEGF with response measurements.
5. Correlate primary tumor tissue VEGF expression with CSF VEGF levels
6. Correlate urine VEGF levels with serum and CSF VEGF levels
7. Evaluate serum and CSF VEGF index

DETAILED DESCRIPTION:
The Study Drug:

Bevacizumab is designed to prevent or slow down the growth of cancer cells by blocking the growth of blood vessels.

Study Drug Administration:

If you are found to be eligible to take part in this study, every 2 weeks, you will receive bevacizumab by vein over about 1 hour.

Study Visits:

At Weeks 2 and 4:

* Samples of CSF from your spinal cord will be collected to check for the presence of cancer cells.
* Blood (about 3 tablespoons) will be drawn for routine tests and to check your blood's ability to clot normally.
* If you already have an Ommaya reservoir tap in place, samples of CSF from your brain will be collected to look for the presence of cancer cells.
* You will be asked about any drugs you may be taking and if you have experienced any side effects.
* You will have a neurological exam.

At Weeks 6, 12, 18, and 24, and then every 8 weeks:

* Samples of CSF from your spinal cord will be collected to check for the presence of cancer cells.
* Blood (about 3 tablespoons) will be drawn for routine tests and to check your blood's ability to clot normally.
* If you already have an Ommaya reservoir tap in place, samples of CSF from your brain will be collected to look for the presence of cancer cells.
* You will have a physical exam (Weeks .
* Your performance status will be recorded.
* You will be asked about any drugs you may be taking and if you have experienced any side effects.
* You will have a neurological exam.
* You will complete the questionnaire about your quality of life.
* You will have an MRI scan to check the status of the disease.
* Urine will be collected to test kidney function and for routine tests. If indicated urine will be collected over a 24 hour period.

Every 2 weeks, your blood pressure will be measured.

Length of Study:

You will be on study for up to 54 weeks (about 1 year). You will be taken off study early if the disease gets worse or you experience intolerable side effects.

End-of-Study Visit:

If you go off study early, the following tests and procedures will be performed:

* You will have a physical exam.
* Your performance status will be recorded.
* You will have a neurological exam.
* Samples of CSF from your spinal cord will be collected to look for the presence of cancer cells.
* Blood (about 3 tablespoons) will be drawn for routine tests and to check your blood's ability to clot normally. You will complete the questionnaire about your quality of life.
* If you already have an Ommaya reservoir tap in place, samples of CSF from your brain will be collected to look for the presence of cancer cells.

Follow-up Visits:

If you do not go off study early, within 4 weeks after the last dose of study drug, every 4 weeks for 3 months, and then every 3 months from then on, you will have follow-up visits. The following tests and procedures will be performed:

* You will have a physical exam.
* Your performance status will be recorded.
* You will have a neurological exam.
* Samples of CSF from your spinal will be collected to look for the presence of cancer cells.
* Blood (about 3 tablespoons) will be drawn for routine tests and to check your blood's ability to clot normally.

You will have an MRI scan to check the status of the disease.

-If you already have an Ommaya reservoir tap in place, samples of CSF from your brain will be collected to look for the presence of cancer cells.

This is an investigational study. Bevacizumab is FDA approved and commercially available for the treatment of colon, breast, and lung cancer. Its use for the treatment of cancer that has spread to the meninges of the brain or the spinal cord is investigational.

Up to 25 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. History of breast cancer, lung cancer or melanoma
2. Diagnosis of NM as proven either by: 1. positive CSF cytology, or 2. magnetic resonance neuro-imaging, or 3. both
3. Age >/=18 years.
4. Routine laboratory studies adequate with bilirubin </= 1.5 x upper limit of normal (ULN), AST < 2.5 x ULN, creatinine <1.0 x ULN, granulocytes >1500, platelets> 75,000; Hb >/= 9.0.
5. Patient able to sign informed consent and willing to participate in study primary objectives
6. At least 1 week from last intrathecal chemotherapy (>2 weeks if liposomal cytarabine). Patients are allowed to have received prior chemotherapy for their tumor. No limit on prior chemotherapies will be made. Patients who have been treated with tyrosine kinase inhibitors are permitted. Prior anti-VEGF targeted therapy is not permitted, unless patient has been off anti-VEGF therapy for 6 months and did not develop NM while on anti-VEGF therapy
7. Karnofsky performance status (KPS) >/= 50%
8. Pre-treatment CSF Indium 111 CSF flow study without evidence of obstruction.
9. Patients on full-dose anticoagulants (e.g., warfarin) with PT international normalized ratio (INR) >1.5 are eligible provided that: 1. Patients are receiving anticoagulation (warfarin or low molecular weight heparins (LMWH)) only if the patients can be off of warfarin for 4-5 days prior to the LP and placed on LMWH in that interim, and if the 'treatment dose' of LMWH can be safely held for 24 hours before and after the LP.
10. ( 9. continued) INR must be <1.2 prior to LP in this circumstance. If patients are receiving thromboprophylaxis dose of LMWH, the patients can be enrolled, but the thromboprophylaxis LMWH must be able to be safely held for 12 hours prior to the LP. 2. The patient has no active bleeding or pathological condition that carries a high risk of bleeding 3. There is no evidence of serious or non-healing wound, ulcer or bone fracture
11. Ventricular reservoir NOT mandatory

Exclusion Criteria:

1. Evidence of active CNS hemorrhage in the brain or tumor lesions
2. Besides NM, other known CNS disease, except for treated brain metastases(Patients must be at least 1 month out from brain irradiation and have no evidence of progression or hemorrhage at that time, as ascertained by clinical examination and brain imaging (MRI or CT) during the screening period). Anticonvulsants (stable dose) are allowed. Treatment for brain metastases may include whole brain radiotherapy, radiosurgery or a combination as deemed appropriate by the treating physician.
3. (2. continued) With respect to irradiation for other purpose (for NM or bone metastases, etc) patients need only 1 week out from the completion of irradiation. Patients with CNS metastases treated by neurosurgical resection or brain biopsy performed within 3 months prior to Day 1 will be excluded.
4. Patients with clinically significant cardiovascular disease are excluded 1) Inadequately controlled HTN (SBP > 140 mmHg and/or diastolic blood pressure (DBP) > 90 mmHg despite antihypertensive medication). 2) Prior history of hypertensive crisis or hypertensive encephalopathy. 3) New York Heart Association (NYHA) Grade II or greater congestive heart failure.
5. ( 4. Continued) 4) History of myocardial infarction or unstable angina within 6 months prior to Day 1. 5) History of stroke or transient ischemic attack within 6 months prior to Day 1. 6) Significant vascular disease (e.g., aortic aneurysm, requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to Day 1. 7) Clinically significant peripheral vascular disease. 8) Serious and inadequately controlled cardiac arrhythmia
6. History of hemoptysis (>/= 1/2 teaspoon of bright red blood per episode) within 1 month prior to Day 1
7. Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
8. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1 or anticipation of need for major surgical procedure during the course of the study
9. Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to Day 1. Ventricular reservoir must have been placed more than 28 days prior to Day 1.
10. History of abdominal fistula or gastrointestinal perforation within 6 months prior to Day 1
11. Serious, non-healing wound, active ulcer, or untreated bone fracture
12. Proteinuria as demonstrated by UPC ratio >/=1.0 at screening or by urine dipstick >/= 2+. (Patients discovered to have >/= 2+ proteinuria on urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate </= 1g of protein in 24 hours to be eligible).
13. Known hypersensitivity to any component of bevacizumab
14. Intrathoracic or extrathoracic lung carcinoma of squamous cell histology. Mixed tumors will be categorized by the predominant cell type unless small cell elements are present, in which case the patient is ineligible; sputum cytology alone is acceptable.
15. (14. continued) Patients with extrathoracic-only squamous cell NSCLC are eligible. Patients with only peripheral lung lesions (of any non squamous NSCLC histology, except small cell histology) will also be eligible (a peripheral lesion is defined as a lesion in which the epicenter of the tumor is </= 2 cm from the costal or diaphragmatic pleura in a three-dimensional orientation based on each lobe of the lung and is >/= 2 cm from the trachea, main, and lobar bronchi).
16. Pregnant (positive pregnancy test) or nursing women. Angiogenesis is critical to fetal development and the inhibition of angiogenesis following administration of AVASTIN is likely to result in adverse effects on pregnancy. There are no adequate and well-controlled studies in pregnant women. Both fertile men and women must agree to use adequate contraceptive measures during study therapy and for at least 2 months after the completion of bevacizumab therapy.
17. General Medical Exclusions 1) Inability to comply with study and/or follow-up procedures 2) Life expectancy of less than 6 weeks 3) Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study other than this Genentech supported study 4) Active malignancy, other than superficial basal cell and superficial squamous (skin) cell, or carcinoma in situ of the cervix within the last 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ivo D. Tremont, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: June 15, 2009 to February 28, 2011. All recruitment done at The University of Texas MD Anderson Cancer Center.
Period: Overall Study
Arm/Group | Bevacizumab
Started | 20
Completed | 13
Not Completed | 7
Not completed — Death | 2
Not completed — Ineligible, Screen Failure | 5

BASELINE CHARACTERISTICS:
Arm/Group | Bevacizumab
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] | 58 [24 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Cerebrospinal Fluid (CSF) Response Rate: Percentage of Participants Positive for Tumor Cells
Description: CSF response for participants with Neoplastic Meningitis (NM) or leptomeningeal disease (LMD) defined as conversion from positive to negative cytology or cytometry as measured routinely by total clearance of malignant cells from the CSF where assessments performed from 2 weeks up to week 54 of treatment. Clearance of malignant cells determined by standard clinical testing using cytospin analysis in clinical laboratory. Percentage reflects number of participants of total treated with no response, e.g. participants with continued positive CSF cytology or flow cytometry.
Time Frame: 1 year (54 weeks) of treatment
Population: Of the 20 registered, 5 were screening failures therefore are not included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 15
percentage of participants | 93

2. Primary Outcome: Median Time to Progression (TTP) and Median Time to Neurological Progression (TTNP)
Description: Time to Progression defined as time to disease progression measured from date of enrollment, confirmation of disease progression via laboratory testing; Time to neurological progression (TTNP) reflects worsening clinical signs/symptoms or development of new clinical signs/symptoms which investigator feels can be attributed to leptomeningeal disease progression and are severe enough to warrant a change in therapy.
Time Frame: 6 weeks
Population: Of the 20 registered, 5 were screening failures therefore are not included in the analysis.
Measure: Median (Full Range); unit: Weeks
Arm/Group | Bevacizumab
Number analyzed (Participants) | 15
Weeks
  TTP | 3 [0 to 6]
  TTNP | 3 [0 to 6]

3. Other Pre Specified Outcome: Participant Response: Cerebrospinal Fluid (CSF) Examination
Description: Neoplastic meningitis is considered an unmeasurable metastatic site by Response Evaluation Criteria in Solid Tumors (RECIST), and as such no standardized methodologies are routinely used; therefore response assessed from cerebrospinal fluid (CSF) obtained via lumbar puncture (and from ventricular reservoir if present) and analyzed for malignant cells along with reference recording of magnetic resonance imaging (MRI) of areas of enhancement over time; however, MRI alone in LMD/NM is considered non-evaluable by RECIST criteria. Those participants with only MRI criteria for enrollment, but who later develop CSF positivity after enrollment were declared "progressors" based on the CSF criteria.
Time Frame: 1 year (54 weeks) of treatment
Population: Of the 20 registered, 5 were screening failures therefore are not included in the analysis.
Measure: Number; unit: participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 15
participants
  No Change/Stable Disease (SD) | 6
  Progressive Disease (PD) | 8
  Complete Remission (CR) | 1

ADVERSE EVENTS:
Time Frame: Adverse event data for study collected for up to 54 weeks (about 1 year), up to 30 days after the date of the last drug administration.
Description: Of the twenty participants, five were not treated and therefore are not included in the adverse event reporting.
Arm/Group | Bevacizumab
Serious Adverse Events (participants affected / at risk) | 11/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab (N=15)
Pain, Gastrointestinal Abdomen (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Wound Complications/Infection (Injury, poisoning and procedural complications) | 1 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Fatique (General disorders) | 1 (1)
Death (General disorders) | 2 (2) — Unrelated to treatment, Disease progression
Seizure (Nervous system disorders) | 3 (3)
Somnolence (Nervous system disorders) | 1 (1)
Nausea/Vomiting (Gastrointestinal disorders) | 1 (1)
Pain, Musculoskeletal (General disorders) | 1 (1)
Confusion (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab (N=15)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 8 (9)
Adult Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 5 (5)
Alkaline phosphatase increased (Investigations) | 4 (6)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 7 (7)
Anorexia (Metabolism and nutrition disorders) | 9 (11)
Anxiety (Psychiatric disorders) | 6 (6)
Aspartate aminotransferase increased (Investigations) | 6 (10)
Ataxia (Nervous system disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (10)
Bilirubin increased (Investigations) | 1 (1)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 3 (5)
Blood glucose increased (Metabolism and nutrition disorders) | 12 (33)
Blood uric acid increased (Metabolism and nutrition disorders) | 2 (6)
Bruising (Injury, poisoning and procedural complications) | 2 (3)
Catheter related infection (Infections and infestations) | 1 (1)
Chest pain (Cardiac disorders) | 2 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 3 (5)
Constipation (Gastrointestinal disorders) | 9 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Creatinine increased (Investigations) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Depressed level of consciousness (Nervous system disorders) | 5 (5)
Depression (Psychiatric disorders) | 6 (7)
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (6)
Diplopia (Eye disorders) | 5 (5)
Dizziness (Nervous system disorders) | 4 (5)
Dry eye syndrome (Eye disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 3 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (7)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Edema limbs (General disorders) | 5 (5)
Facial muscle weakness (Nervous system disorders) | 2 (2)
Facial nerve disorder (Nervous system disorders) | 1 (2)
Fatigue (General disorders) | 15 (23)
Fecal incontinence (Gastrointestinal disorders) | 2 (2)
Fever (General disorders) | 2 (2)
Gait abnormal (Musculoskeletal and connective tissue disorders) | 13 (17)
Gastrointestinal (Other) (Gastrointestinal disorders) | 3 (3)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 8 (13)
Hearing loss (Ear and labyrinth disorders) | 3 (3)
Hemoglobin decreased (Investigations) | 11 (34)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 3 (4)
Hypotension (Vascular disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infection (Infections and infestations) | 2 (2)
Insomnia (Psychiatric disorders) | 10 (10)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Keratitis (Eye disorders) | 1 (1)
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 9 (16)
Lymphatics (Other) (Blood and lymphatic system disorders) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 11 (37)
Memory impairment (Nervous system disorders) | 4 (4)
Metabolic/Laboratory (Other) (Metabolism and nutrition disorders) | 15 (55)
Mini mental status examination abnormal (Psychiatric disorders) | 1 (1)
Mucositis oral (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 7 (10)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 3 (5)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 7 (10)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (2)
Musculoskeletal (Other) (Musculoskeletal and connective tissue disorders) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 12 (21)
Neurology (Other) (Nervous system disorders) | 9 (12)
Neutrophil count decreased (Blood and lymphatic system disorders) | 3 (5)
Ocular/Visual (Other) (Eye disorders) | 3 (3)
Optic nerve disorder (Eye disorders) | 1 (1)
Pain (General disorders) | 3 (3)
Pain (Other) (General disorders) | 4 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (13)
Palpitations (Cardiac disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 7 (9)
Platelet count decreased (Investigations) | 4 (4)
Pneumonia (Infections and infestations) | 1 (1)
Pulmonary (Other) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pyramidal tract syndrome (Nervous system disorders) | 3 (3)
Rash desquamating (Skin and subcutaneous tissue disorders) | 2 (3)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Seizure (Nervous system disorders) | 3 (4)
Sepsis (Infections and infestations) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 6 (6)
Serum cacium decreased (Metabolism and nutrition disorders) | 5 (13)
Serum cholesterol increased (Metabolism and nutrition disorders) | 1 (1)
Serum glucose decrease (Metabolism and nutrition disorders) | 2 (5)
Serum magnesium decreased (Metabolism and nutrition disorders) | 6 (10)
Serum phosphate decreased (Metabolism and nutrition disorders) | 2 (4)
Serum potassium increased (Metabolism and nutrition disorders) | 1 (2)
Serum sodium decreased (Metabolism and nutrition disorders) | 8 (18)
Serum sodium increased (Metabolism and nutrition disorders) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 7 (14)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Speech disorder (Nervous system disorders) | 5 (6)
Syncope (Nervous system disorders) | 1 (1)
Syncope vasovagal (Nervous system disorders) | 1 (1)
Taste alteration (Nervous system disorders) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Tremor (Nervous system disorders) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 3 (3)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 3 (4)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Vision blurred (Eye disorders) | 4 (4)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 10 (14)
Weight gain (Investigations) | 1 (1)
Weight loss (Investigations) | 4 (7)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes